CLINICAL TRIAL: NCT07302542
Title: Impact of Oat Milk Consumption on Gastrointestinal Transit and Defecation Frequency: A Controlled Intervention Trial in Adults
Brief Title: Oat Milk for Laxation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Xiuwen Ren, Doctoral Student, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MNCGJH-20250903-0022
Record Dates: First submitted 2025-11-30; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Dietary Supplement: oat milk
- Control Group (No Intervention)

INTERVENTIONS:
Dietary Supplement: oat milk — The intervention group will consume 250 mL of Mengniu Daily Fiber Oat Milk daily for 28 consecutive days
  Arms: Intervention Group

SUMMARY:
This study intends to recruit 90-100 constipated participants aged 25-50 years, including an equal number of males and females, from the faculty and logistics staff of Capital Medical University. Participants will be randomly divided into an intervention group (55-60 individuals) and a control group (35-40 individuals). The intervention group will consume 250 mL of Mengniu Daily Fiber Oat Milk daily for 4 weeks, while the control group will not receive oat milk intervention. Both groups will maintain their original lifestyles, including diet, sleep, and exercise, throughout the study period. Baseline surveys, dietary surveys, blood and urine routine tests, blood biochemical indices, and intestinal flora detection will be conducted before and after the intervention. Defecation status will be recorded, and gastrointestinal symptoms will be assessed using a Gastrointestinal Symptom Rating Scale. Statistical analysis will be performed to determine the laxative efficacy of oat milk.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of non-organic and habitual constipation;

Reduced defecation frequency;

Increased stool hardness;

Fewer than 4 bowel movements per week;

Exclusion Criteria:

Inability to take food orally or inability to comply with the required intake of the test product;

Known allergy to oats or related products;

Unclear primary gastrointestinal complaints;

Physical weakness that prevents participation in the trial;

History of surgery within the past 30 days that may cause constipation；

Recent constipation caused by severe organic gastrointestinal lesions (e.g., colon cancer, severe enteritis, intestinal obstruction, inflammatory bowel disease);

Constipation accompanied by significant abdominal pain;

Acute gastrointestinal diseases within the past 30 days;

Severe systemic diseases involving the cardiovascular, hepatic, renal, or hematopoietic systems;

Ongoing treatment for comorbid conditions that may interfere with study participation;

Recent use of substances related to the tested function that may influence outcome measurements.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Changes in Intestinal Flora Composition Assessed by Metagenomic Sequencing | Collect feces and evaluate at baseline and at the fourth week.
  Fecal samples from a randomly selected subgroup (30 participants in the intervention group and 15 in the control group) will be collected before and after the intervention. Metagenomic sequencing will be used to evaluate changes in intestinal microbiota composition and functional gene pathways, including metabolism-, immunity-, and disease-related gene sets. This outcome explores potential mechanisms by which the intervention exerts laxative effects.

SECONDARY OUTCOMES:
Changes in Gastrointestinal Symptoms Assessed by the Gastrointestinal Symptom Rating Scale | Participates will fill out the questionnaire at baseline, Week 2, and Week 4.
  Gastrointestinal symptoms will be evaluated using the Gastrointestinal Symptom Rating Scale (GSRS, 15 items; score range: 1-7, with higher scores indicating more severe symptoms). Assessments will be conducted at baseline, Week 2, and Week 4. Symptoms include reflux, abdominal pain, indigestion, diarrhea, and constipation.

IPD SHARING:
Plan to Share IPD: No